CLINICAL TRIAL: NCT03848572
Title: A Randomized Study of Repetitive Assessement of PRECISE-DAPT Score During Dual Antiplatelet Therapy: The RE-SCORE Trial
Brief Title: Repetitive Assessement of PRECISE-DAPT Score
Acronym: RE-SCORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Assistant Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019/D/101
Record Dates: First submitted 2019-02-19; First posted 2019-02-20 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Cardiovascular Diseases; Interventional Cardiology
Keywords: Dual Anti-platelet Therapy; Bleeding
MeSH Terms: conditions — Cardiovascular Diseases; Hemorrhage

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Patients will enter standard 12-month clinical follow-up
- Re-Score strategy (Experimental): Patients will enter a novel strategy of 12-month follow with repetitive assessment of PRECISE-DAPT score at 3-month intervals
  Interventions: Diagnostic Test: Repetitive assessment of PRECISE-DAPT score

INTERVENTIONS:
Diagnostic Test: Repetitive assessment of PRECISE-DAPT score — The PRECISE-DAPT score, which takes into consideration age, creatinine clearance, haemoglobin, white blood-cell count and previous spontaneous bleeding, will be reassessed every 3 months during the 12-month follow-up period
  Arms: Re-Score strategy

SUMMARY:
Patients treated with percutaneous coronary intervention (PCI) require dual antiplatelet therapy (DAPT). Preliminary assessment of the PRECISE-DAPT score is mandatory in order to assess the risk of bleeding while on DAPT. The score takes into consideration age, creatinine clearance, haemoglobin, white blood- cell count and previous spontaneous bleeding. One should consider, however, that some of the variables included in the PRECISE-DAPT score might change with time. As a consequence, the PRECISE-DAPT score should not be considered a static score as it might vary after the initial computation.

It remains unknown, however, if the use of the delta PRECISE-SCORE, which reflects the change in score between baseline and follow-up, might help to improve the management of PCI patients in order to decrease the bleeding risk during follow-up.

DETAILED DESCRIPTION:
The RE-SCORE trial is a multicenter study aimed at comparing usual care of patients treated with PCI with a novel strategy of change of therapy during follow-up on the base of the Delta PRECISE-DAPT score, as assessed every 3 months in PCI patients receiving DAPT. The primary end-point of the study is the occurrence of bleeding, as defined according to the criteria of the Bleeding Academic Research Consortium (BARC). The second end-point is a composite of cardiac death, myocardial infarction, stroke, definite or probable stent thrombosis (ST), or BARC criteria type 2, 3 or 5 bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients undergoing percutaneous coronary intervention
* Indication to dual antiplatelet therapy for at least 3 months

Exclusion Criteria:

- Contraindications to dual antiplatelet therapy lasting more than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Bleeding episode | 12 months
  The time to first occurrence of clinically relevant bleeding, defined as Bleeding Academic Research Consortium (BARC) Types 2, 3 or 5 bleeding

SECONDARY OUTCOMES:
Ischemic episode | 12 months
  The time to first occurrence of cardiovascular death, non-fatal myocardial infarction, ischemic stroke or ischemia-driven revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Gaudio, MD, Study Chair — Sapienza University
Locations (2):
- Italy (2):
  - San Raffaele Pisana, Rome
  - Sapienza University, Rome

IPD SHARING:
Plan to Share IPD: No